CLINICAL TRIAL: NCT06466421
Title: Clinical Study to Compare The Safety and Possible Efficacy of Fexofenadine Versus Gabapentin for Uremic Pruritus in Patients on Regular Hemodialysis
Brief Title: Fexofenadine Versus Gabapentin for Uremic Pruritus in Patients on Regular Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Ihab Hosny Mohamed Elfalaha, Pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Fexof vs Gaba for UP in RHD
Record Dates: First submitted 2024-06-07; First posted 2024-06-20 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Uremic Pruritus; Chronic Kidney Disease-associated Pruritus; Hemodialysis; End-stage Renal Disease; Renal Replacement Therapy; ESRD
Keywords: pruritus; Hemodialysis; ESRD; RHD; Fexofenadine; Gabapentin; Interleukin 6; IL-6; Substance P; SP; CKD-aP; Chronic Kidney Disease-associated Pruritus; Uremic; UP; Uremic Pruritus; End-stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic; Pruritus | interventions — fexofenadine; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: (Gabapentin group) (Active Comparator): 30 patients will receive Gabapentin 100 mg after each dialysis session (thrice weekly). Dose may be titrated after 2 weeks, according to response and tolerability, to 100 mg orally once daily for 3 months.
  Interventions: Drug: Gabapentin
- Group 2: (Fexofenadine group) (Experimental): 30 patients will receive Fexofenadine 60 mg orally once daily for 3 months.
  Interventions: Drug: Fexofenadine

INTERVENTIONS:
Drug: Fexofenadine — Fexofenadine 60 mg orally once daily for 3 months
  Arms: Group 2: (Fexofenadine group)
Drug: Gabapentin — 100 mg after each dialysis session (thrice weekly). Dose may be titrated after 2 weeks, according to response and tolerability, to 100 mg orally once daily for 3 months.
  Arms: Group 1: (Gabapentin group)

SUMMARY:
Several studies investigated the effectiveness of Gabapentin in Uremic Pruritus (UP). No previous studies investigated the use of fexofenadine in UP. The aim of this trial is to assess the safety and possible efficacy of fexofenadine in patients with UP.

DETAILED DESCRIPTION:
A randomized controlled single center parallel study, that will recruit 60 participants with end stage renal disease (ESRD) on regular hemodialysis (RHD) with uremic pruritus (UP). Patients will be randomized to either Fexofenadine (60 mg orally once daily), or Gabapentin (100 mg orally after each dialysis session, "thrice weekly", with titration according to response to 100 mg orally once daily). Participants will continue treatment for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* ESRD on regular hemodialysis.
* Moderate and severe Uremic Pruritus as assessed by Visual Analogue Scale.
* Able to provide an informed consent.

Exclusion Criteria:

* Age < 18 years old.
* Patients not on regular hemodialysis.
* Pruritus due to other cause.
* Cancer patients.
* Pregnancy or breastfeeding.
* Patients with history of substance abuse.
* Patients with myasthenia gravis.
* Patients who refuse or are unable to provide an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
The Visual Analogue Scale (VAS) | 3 months
  The change in mean score of Visual Analogue Scale (VAS) from baseline.
Skindex score | 3 months
  The change in mean Skindex score from baseline.
Kidney Disease Quality of Life Short Form (KDQOL-SF™) | 3 months
  The change in mean KDQOL-SF score from baseline.

SECONDARY OUTCOMES:
Interleukin-6 (IL-6) | 3 months
  The change in mean serum level of Interleukin-6 (IL-6) from baseline.
Substance P | 3 months
  The change in mean serum level of Substance P from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Sahar M El-Haggar, PhD, Study Chair — Tanta University; Ahmed M Hussein, PhD, Study Director — Helwan University; Mohamed I Hosney, PharmD, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yosipovitch G, Rosen JD, Hashimoto T. Itch: From mechanism to (novel) therapeutic approaches. J Allergy Clin Immunol. 2018 Nov;142(5):1375-1390. doi: 10.1016/j.jaci.2018.09.005. PMID 30409247
- [Background] Verduzco HA, Shirazian S. CKD-Associated Pruritus: New Insights Into Diagnosis, Pathogenesis, and Management. Kidney Int Rep. 2020 May 8;5(9):1387-1402. doi: 10.1016/j.ekir.2020.04.027. eCollection 2020 Sep. PMID 32954065
- [Background] Sukul N, Speyer E, Tu C, Bieber BA, Li Y, Lopes AA, Asahi K, Mariani L, Laville M, Rayner HC, Stengel B, Robinson BM, Pisoni RL; CKDopps and CKD-REIN investigators. Pruritus and Patient Reported Outcomes in Non-Dialysis CKD. Clin J Am Soc Nephrol. 2019 May 7;14(5):673-681. doi: 10.2215/CJN.09600818. Epub 2019 Apr 11. PMID 30975656
- [Background] Smith BH, Higgins C, Baldacchino A, Kidd B, Bannister J. Substance misuse of gabapentin. Br J Gen Pract. 2012 Aug;62(601):406-7. doi: 10.3399/bjgp12X653516. No abstract available. PMID 22867659
- [Background] Schricker S, Heider T, Schanz M, Dippon J, Alscher MD, Weiss H, Mettang T, Kimmel M. Strong Associations Between Inflammation, Pruritus and Mental Health in Dialysis Patients. Acta Derm Venereol. 2019 May 1;99(6):524-529. doi: 10.2340/00015555-3128. PMID 30673107
- [Background] Ricardo AC, Hacker E, Lora CM, Ackerson L, DeSalvo KB, Go A, Kusek JW, Nessel L, Ojo A, Townsend RR, Xie D, Ferrans CE, Lash JP; CRIC Investigators. Validation of the Kidney Disease Quality of Life Short Form 36 (KDQOL-36) US Spanish and English versions in a cohort of Hispanics with chronic kidney disease. Ethn Dis. 2013 Spring;23(2):202-9. PMID 23530302
- [Background] Park IH, Um JY, Cho JS, Lee SH, Lee SH, Lee HM. Histamine Promotes the Release of Interleukin-6 via the H1R/p38 and NF-kappaB Pathways in Nasal Fibroblasts. Allergy Asthma Immunol Res. 2014 Nov;6(6):567-72. doi: 10.4168/aair.2014.6.6.567. Epub 2014 Jul 28. PMID 25374757
- [Background] Oweis AO, Al-Qarqaz F, Bodoor K, Heis L, Alfaqih MA, Almomani R, Obeidat MA, Alshelleh SA. Elevated interleukin 31 serum levels in hemodialysis patients are associated with uremic pruritus. Cytokine. 2021 Feb;138:155369. doi: 10.1016/j.cyto.2020.155369. Epub 2020 Nov 19. PMID 33221158
- [Background] Oh G, Moga DC, Fardo DW, Abner EL. The association of gabapentin initiation and neurocognitive changes in older adults with normal cognition. Front Pharmacol. 2022 Nov 25;13:910719. doi: 10.3389/fphar.2022.910719. eCollection 2022. PMID 36506564
- [Background] Gobo-Oliveira M, Pigari VG, Ogata MS, Miot HA, Ponce D, Abbade LP. Gabapentin versus dexchlorpheniramine as treatment for uremic pruritus: a randomised controlled trial. Eur J Dermatol. 2018 Aug 1;28(4):488-495. doi: 10.1684/ejd.2018.3356. PMID 29976533
- [Background] Fehrenbacher JC, Taylor CP, Vasko MR. Pregabalin and gabapentin reduce release of substance P and CGRP from rat spinal tissues only after inflammation or activation of protein kinase C. Pain. 2003 Sep;105(1-2):133-41. doi: 10.1016/s0304-3959(03)00173-8. PMID 14499429
- [Background] Elman S, Hynan LS, Gabriel V, Mayo MJ. The 5-D itch scale: a new measure of pruritus. Br J Dermatol. 2010 Mar;162(3):587-93. doi: 10.1111/j.1365-2133.2009.09586.x. Epub 2009 Dec 1. PMID 19995367
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Background] Davidson S, Giesler GJ. The multiple pathways for itch and their interactions with pain. Trends Neurosci. 2010 Dec;33(12):550-8. doi: 10.1016/j.tins.2010.09.002. Epub 2010 Nov 5. PMID 21056479
- [Background] Chren MM, Lasek RJ, Quinn LM, Mostow EN, Zyzanski SJ. Skindex, a quality-of-life measure for patients with skin disease: reliability, validity, and responsiveness. J Invest Dermatol. 1996 Nov;107(5):707-13. doi: 10.1111/1523-1747.ep12365600. PMID 8875954
- [Background] Ningombam A, Handa S, Srivastava N, Mahajan R, De D. Addition of oral fexofenadine to topical therapy leads to a significantly greater reduction in the serum interleukin-31 levels in mild to moderate paediatric atopic dermatitis. Clin Exp Dermatol. 2022 Apr;47(4):724-729. doi: 10.1111/ced.15032. Epub 2022 Jan 6. PMID 34826148